CLINICAL TRIAL: NCT06913777
Title: An Open-Label, Multicenter, Randomized Controlled Phase III Clinical Study of Neoadjuvant Chemotherapy Based on SNF Classification With or Without Precision Medicine Agents for Early-Stage or Locally Advanced HR+/HER2- Breast Cancer
Brief Title: Neoadjuvant SNF Precision Therapy Phase III
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Director of General Surgery of Fudan Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N090
Record Dates: First submitted 2025-03-30; First posted 2025-04-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Neoadjuvant Therapy
MeSH Terms: interventions — famitinib; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): chemotherapy (wP-EC）
  Interventions: Drug: Chemotherapy (wP-EC)
- Precision group (Experimental): chemotherapy + target therapy
  Interventions: Drug: Targeted therapy agents: SNF2 -adebrelimab + famitinib; SNF3 -fluzoparib; SNF4 -apatinib; Drug: Chemotherapy (wP-EC)

INTERVENTIONS:
Drug: Targeted therapy agents: SNF2 -adebrelimab + famitinib; SNF3 -fluzoparib; SNF4 -apatinib — The backbone is chemotherapy which will be used in the control group. The precision group will add targeted therapy agents which were determined according to SNF classification: the SNF2 subtype add adebrelimab combined with famitinib, the SNF3 subtype receives fluzoparib, and the SNF4 subtype receives apatinib.
  Arms: Precision group
Drug: Chemotherapy (wP-EC) — Chemotherapy : weely nab-P * 12- EC * 4

SUMMARY:
This study is a prospective, open-label, multicenter, randomized controlled Phase III clinical trial designed to compare the efficacy and safety of neoadjuvant chemotherapy based on SNF classification with or without precision medicine agents in previously untreated patients with early-stage or locally advanced HR+/HER2- breast cancer.

ELIGIBILITY:
Eligibility Criteria:

1. Female patients aged 18 to 70 years.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
3. Histologically confirmed HR-positive/HER2-negative breast cancer (defined as: (1) ER-positive: ≥10% tumor cells positive by immunohistochemistry (IHC).

(2) PR-positive: ≥10% tumor cells positive by IHC. (3) HR-positive: ER and/or PR positive. (4) HER2-negative: HER2 0-1+ by IHC or HER2 2+ with negative FISH (no amplification).

4. Confirmed SNF2/3/4 subtype based on H&E staining combined with digital pathology molecular subtyping.

5. Clinical tumor stage: cT1c-T2, cN1-N2 or cT3-T4, cN0-N2. 6. Agreement to undergo breast cancer surgery if meeting the criteria for resection after neoadjuvant therapy.

7. Adequate organ function, meeting the following criteria: Hemoglobin (Hb) ≥90 g/L; Absolute neutrophil count (ANC) ≥1.5×10⁹/L; Platelet count (PLT) ≥75×10⁹/L; Total bilirubin (TBIL) ≤1.5×ULN (upper limit of normal); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3×ULN; Serum creatinine (Cr) ≤1×ULN; Creatinine clearance rate (CrCl) >50 mL/min (calculated by Cockcroft-Gault formula).

8. Baseline left ventricular ejection fraction (LVEF) ≥55% measured by echocardiography or MUGA scan.

9. Negative serum pregnancy test for women of childbearing potential. Contraception requirement: Women of childbearing potential must use medically approved contraception during treatment and for at least 3 months after the last dose of the study drug.

10Voluntary participation with signed informed consent, good compliance, and willingness to follow up.

Exclusion Criteria:

1. Stage IV (metastatic) breast cancer.
2. History of invasive breast cancer.
3. History of ductal carcinoma in situ (DCIS) or lobular carcinoma in situ (LCIS).
4. Prior systemic therapy for breast cancer (chemotherapy, endocrine therapy, or anti-HER2 therapy), or prior excisional biopsy/radiotherapy of primary breast tumor and/or axillary lymph nodes (excluding diagnostic biopsy for primary breast cancer or surgery for benign breast tumors).
5. Other malignancies within the past 5 years (except cured cervical carcinoma in situ or non-melanoma skin cancer).
6. Participation in any other investigational drug study within 4 weeks prior to randomization.
7. Peripheral neuropathy ≥ Grade 2 (per NCI-CTCAE v5.0).
8. Severe cardiovascular or cerebrovascular diseases within 6 months prior to randomization, including but not limited to:

   * Congestive heart failure,
   * Unstable angina,
   * Severe uncontrolled arrhythmias,
   * Clinically significant valvular disease,
   * Uncontrolled severe hypertension,
   * Myocardial infarction, or
   * Cerebrovascular accident.
9. Any severe uncontrolled systemic disease that may interfere with the treatment plan, including significant cardiovascular, pulmonary, or metabolic disorders.
10. Major surgery within 4 weeks prior to randomization without full recovery, or anticipated need for major surgery during the study treatment.
11. Systemic corticosteroid use (>10 mg prednisone equivalent daily) or other immunosuppressants within 2 weeks prior to the first dose of study drug (except for prophylactic anti-allergy or antiemetic purposes).

    * Inhaled/topical steroids or physiologic steroid replacement doses (≤10 mg/day prednisone equivalent) are permitted in the absence of active autoimmune disease.
12. Administration of anti-cancer vaccines or live vaccines within 4 weeks prior to the first dose of study drug.
13. Active autoimmune disease or history of autoimmune disorders (e.g., interstitial lung disease, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyper/hypothyroidism), EXCEPT:

    * Vitiligo,
    * Childhood asthma/allergies resolved without intervention in adulthood,
    * Stable hypothyroidism on hormone replacement,
    * Type 1 diabetes on stable insulin therapy.
    * Exclusion: Asthma requiring bronchodilators.
14. Immunodeficiency (e.g., HIV-positive, congenital/acquired immune deficiency) or history of organ/allogeneic bone marrow transplantation.
15. History of interstitial lung disease (except radiation pneumonitis without steroid treatment) or non-infectious pneumonitis.
16. Active liver disease, including:

    * Hepatitis B (HBsAg-positive with HBV-DNA ≥1000 IU/mL),
    * Hepatitis C (HCV-Ab-positive with detectable HCV-RNA), or
    * Autoimmune hepatitis.
17. Pregnancy or lactation.
18. Known hypersensitivity to the study drug(s), its excipients, or severe allergic reactions to monoclonal antibodies.
19. History of substance abuse, alcoholism, or drug addiction.
20. Uncontrolled psychiatric/neurological disorders (e.g., epilepsy, dementia) or poor compliance.
21. Any other condition that may increase study risk, interfere with treatment/outcomes, or render the patient unsuitable for participation per investigator's judgment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate using the definition of ypT0/Tis ypN0 ((i.e., no invasive residual in breast or nodes; noninvasive breast residuals allowed) at the time of definitive surgery) | Up to approximately 1 year
  pCR rate after neoadjuvant treatment, defined as the proportion of participants who have no evidence by H&E staining of residual invasive disease in the complete resected breast specimen and all sampled regional lymph nodes (ypT0/Tis ypN0) by investigator assessment following completion of neoadjuvant therapy.

SECONDARY OUTCOMES:
Event-free survival (EFS) rate at 12, 24, 36-month | Up to approximately 3 years
  EFS is defined as time from date of randomisation until disease progression precluding initial surgery, invasive disease recurrence (local, regional, distant, or contralateral), or death from any cause.
Invasive disease-free survival (IDFS) rate at 12, 24, 36-month | Up to approximately 3 years
  IDFS is defined as time from surgery until invasive disease recurrence (local, regional, distant, or contralateral), or death from any cause.
Overall Survival (OS) | Approximately 5 years
  OS is defined as the time from randomisation until the date of death due to any cause.
Objective Response Rate (ORR) | Approximately 1 year
  ORR is defined as the proportion of participants who have a complete response (CR) or partial response (PR) based on BICR and investigator assessment using RECIST 1.1.
Safety including adverse events (AEs), severe adverse events (SAEs) and adverse events of special interest (AESI). | Up to approximately 1.5 years
  Incidence of AEs, SAE, AESIs (interstitial lung disease, LVEF decrease), AEs resulting in study intervention interruption and discontinuation, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No